CLINICAL TRIAL: NCT00800033
Title: Effectiveness of Pulse-Based Foods Combined With Exercise for Improving Components of the Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PRO0822
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; lipids; blood pressure; body composition
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aerobic exercise training (Experimental)
  Interventions: Behavioral: Aerobic exercise training
- Resistance exercise training (Placebo Comparator)
  Interventions: Behavioral: Aerobic exercise training
- pulse diet (Experimental): Pulse based diet containing peas, lentils, and beans
  Interventions: Dietary Supplement: pulse based diet
- Regular diet (No Intervention)

INTERVENTIONS:
Behavioral: Aerobic exercise training — Walking, jogging, rowing, cycling to be done 5 times per week for 45 minutes per session (3 supervised sessions, 2 sessions at home) for 5 months
  Arms: Aerobic exercise training; Resistance exercise training
Dietary Supplement: pulse based diet — Two pulse-based meals per day (lentils, beans, chickpeas, or peas) for 2 months, followed by 1-month washout and then a normal diet for 2 months (order of diets is randomized)
  Arms: pulse diet

SUMMARY:
The investigators specific objective is to determine the effectiveness of a pulse-based diet combined with an exercise training program for reducing the risk of metabolic syndrome in older adults. The metabolic syndrome is a cluster of risk factors that predispose one to the development of diabetes and cardiovascular disease. These risk factors include increased abdominal obesity, high blood triglyceride levels, low blood high-density lipoproteins, high blood pressure, high blood glucose and insulin levels, and increased inflammation. The investigators hypothesize that a pulse-based diet combined with exercise training will be very effective for reducing the risks of the metabolic syndrome because each intervention acts on different components of the metabolic syndrome.

The design will involve a randomized single-blind cross-over for the pulse-based diet, and a single blind randomized parallel group assignment for the exercise-based intervention. 100 subjects will be randomized to receive the pulse-based diet or their regular diet for 2 months and then cross-over to receive the opposite diet for 2 months, separated by a one-month "wash out". Subjects will be further randomized to exercise or "exercise placebo" groups for the duration of the trial (i.e. 5 months). The exercise intervention will involve aerobic training as this is most effective for reducing metabolic syndrome risk.

Dependent variables will be measured at 4 time points: baseline, after the first 2-month diet, before the second 2-month diet (i.e. after the washout) and at the end of the second 2-month diet. These variables will include: Serum triglycerides, high density lipoproteins, C-reactive protein (as an inflammatory marker), glucose, and insulin, trunk body fat, and blood pressure. A composite metabolic syndrome score will be determined by converting each of these variables into Z-scores and determining the mean of these Z-scores. Secondary variables will include other serum lipids, including low density lipoproteins and total cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* men and women over the age of 50y

Exclusion Criteria:

* allergies to beans, peas, lentils, chickpeas
* currently taking medication for blood lipids
* currently engaged in vigorous aerobic activity greater than 2 times per week

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome score | baseline, 2 months, 3 months, 5 months

SECONDARY OUTCOMES:
Plasma glucose | baseline, 2 months, 3 months, 5 months
Plasma insulin | baseline, 2 months, 3 months, 5 months
High density lipoproteins | baseline, 2 months, 3 months, 5 months
Triacylglycerol | baseline, 2 months, 3 months, 5 months
Waist circumference | baseline, 2 months, 3 months, 5 months
C-reactive protein | baseline, 2 months, 3 months, 5 months
Lean body mass | baseline, 2 months, 3 months, 5 months
Fat mass | baseline, 2 months, 3 months, 5 months
Whole body bone mineral | baseline, 2 months, 3 months, 5 months
Hip bone mineral | baseline, 2 months, 3 months, 5 months
Lumbar spine bone mineral | baseline, 2 months, 3 months, 5 months
Low density lipoproteins | baseline, 2 months, 3 months, 5 months
Total cholesterol | baseline, 2 months, 3 months, 5 months
Blood Pressure | baseline, 2 months, 3 months, 5 months
Aerobic fitness - modified Canadian Test of Fitness | baseline, 2 months, 3 months, 5 months
Strength | baseline, 2 months, 3 months, 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip D Chilibeck, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan, Canada